CLINICAL TRIAL: NCT06002971
Title: Validation of the CONNEQT Blood Pressure Monitoring System in a Pregnant Patient Population
Brief Title: CONNEQT Pulse Validation Study
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit intended patient population
Sponsor: Mount Carmel Health System (Other)
Collaborators: AtCor Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Robin Driver, Principal Investigator, Mount Carmel Health System
Other Study IDs: 230608-6
Record Dates: First submitted 2023-08-08; First posted 2023-08-21 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-10

CONDITIONS: Pregnancy Related; Pre-Eclampsia; Gestational Hypertension
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced | interventions — Blood Pressure Determination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Normotensive: Normotensive pregnant patients beyond the first trimester with systolic blood pressure <140 mmHg and diastolic blood pressure <90 mmHg
  Interventions: Device: Blood pressure measurement
- Hypertensive: Hypertensive pregnant patients beyond the first trimester:
  i) without proteinuria >300 mg in 24 h; and ii) with systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥ 90 mmHg
  Interventions: Device: Blood pressure measurement
- Pre-Eclampsia: Pre-eclampsia patients beyond the first trimester:
  i) with proteinuria >300 mg in 24 h; and ii) with systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥ 90 mmHg
  Interventions: Device: Blood pressure measurement

INTERVENTIONS:
Device: Blood pressure measurement — Serial blood pressure measurements to compare reference auscultatory sphygmomanometer to CONNEQT Pulse according to ISO 81060-2.

SUMMARY:
The purpose of this study is to validate the accuracy of the CONNEQT Pulse blood pressure monitoring system for the measurement of blood pressure as compared to a gold standard, auscultatory sphygmomanometer in a pregnant population.

DETAILED DESCRIPTION:
Clinical staff will review patient's medical record to determine eligibility. Following informed consent, a brief medical history will be collected. Serial blood pressure measurements will be collected to compare an auscultatory sphygmomanometer to blood pressure measurements of the CONNEQT Pulse blood pressure monitoring system in a pregnant population according to ISO protocol 81060-2.

ELIGIBILITY:
All Groups:

1. Able to provide informed consent
2. Pregnant patient, beyond the first trimester (greater than 12 weeks of gestation)
3. 18 years of age, or older

Normotensive:

1. Systolic blood pressure <140 mmHg (18,66 kPa) and diastolic blood pressure <90 mmHg (12 kPa)

Hypertensive:

1. Without proteinuria >300 mg in 24 h; and
2. With systolic blood pressure ≥140 mmHg (18,66 kPa) or diastolic blood pressure ≥ 90 mmHg (12 kPa)

Pre-Eclampsia:

1. With proteinuria >300 mg in 24 h; and
2. With systolic blood pressure ≥140 mmHg (18,66 kPa) or diastolic blood pressure ≥ 90 mmHg (12,00 kPa)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant patients 18 years or older and beyond the first trimester, as defined as 12 completed weeks of gestation.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Comparison of reference auscultatory blood pressure readings to CONNEQT Pulse blood pressure readings. | Up to 60 minutes
  Paired means and standard deviations of both systolic and diastolic blood pressure readings will be analyzed according to section 5.2.4.1.2 of ISO 81060-2 protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Carmel East, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No